CLINICAL TRIAL: NCT02923531
Title: A Phase 1B/2A Trial Adding X4P-001 in Patients Receiving Nivolumab for Treatment of Advanced Clear Cell Renal Cell Carcinoma
Brief Title: Addition of X4P-001 to Nivolumab Treatment in Participants With Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to low enrollment, the study was terminated early.
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X4P-001-RCCB
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-11

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — mavorixafor; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- X4P-001 Plus Nivolumab (Experimental): Participants will receive X4P-001 400 milligrams (mg) (as 4 capsules of 100 mg each) orally once daily in combination with nivolumab 240 mg intravenous (IV) infusion (over 60 minutes) every 2 weeks. Study medication will be administered in 28-day cycles and will continue until treatment-limiting toxicity or disease progression.
  Interventions: Drug: X4P-001; Drug: Nivolumab

INTERVENTIONS:
Drug: X4P-001 — X4P-001 will be administered as per the dose and schedule specified in the arm.
Drug: Nivolumab — Nivolumab will be administered as per the dose and schedule specified in the arm.
  Other Names: Opdivo

SUMMARY:
The purpose of this study is to determine if the combination of X4P-001 plus nivolumab is safe and tolerable. Secondly, the study will investigate if adding X4P-001 to nivolumab treatment has an effect on the body and the cancer tumor, in participants receiving nivolumab but not exhibiting a radiological response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of Renal Cell Carcinoma with a documented clear cell component (ccRCC).
* Currently receiving nivolumab and considered by Investigator to have the potential to derive clinical benefit from continuing treatment with nivolumab.
* Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria on current nivolumab treatment (prior to initiation of this study), has a best response of confirmed stable disease (SD) or confirmed progressive disease (PD). Confirmed SD or confirmed PD refers to a response that is confirmed by a second scan which is at least 4 weeks apart from the previous scan.
* At least one extra-renal measurable target lesion meeting the criteria of RECIST Version 1.1.
* Agree to use contraception from screening, through the study, and for at least 5 months after the last dose of nivolumab as follows: for women of childbearing potential agree to use highly-effective contraceptive methods; for males, agree to use a condom with sexual partner.

Exclusion Criteria:

* Pregnant or nursing.
* Life expectancy of less than 3 months.
* Performance status greater than or equal to (≥) 2 (Eastern Cooperative Oncology Group [ECOG] criteria).
* New York Heart Association (NYHA) Class III or IV, uncontrolled hypertension, or clinically significant arrhythmia.
* Previously received X4P-001.
* Has a second malignancy. Except: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type.
* Has active central nervous system (CNS) metastases (including evidence of cerebral edema by Magnetic Resonance Imaging [MRI], or progression from prior imaging study, or any requirement for steroids, or clinical symptoms of/from CNS metastases) within 28 days prior to study treatment. Subjects with known CNS metastases must have a baseline MRI scan within 28 days of study treatment.
* Ongoing clinical adverse events National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade greater than (>) 2 resulting from prior cancer therapies.
* Known history of Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS); or positive test for hepatitis C virus (HCV), or hepatitis B surface antigen (HBsAg).
* History of clinically significant or uncontrolled cardiac, hepatic, or pulmonary disease.
* Has had within the past 6 months the occurrence of one or more of the following events: myocardial infarction, cerebrovascular accident, deep vein thrombosis, pulmonary embolism, hemorrhage (NCI CTCAE Grade 3 or 4), chronic liver disease (meeting criteria for Child-Pugh Class B or C), or organ transplantation.
* Inadequate hematologic, hepatic, or renal function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — X4 Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Washington D.C., District of Columbia
  - Boston, Massachusetts
  - Hackensack, New Jersey
  - Chapel Hill, North Carolina

REFERENCES:
- [Derived] Choueiri TK, Atkins MB, Rose TL, Alter RS, Ju Y, Niland K, Wang Y, Arbeit R, Parasuraman S, Gan L, McDermott DF. A phase 1b trial of the CXCR4 inhibitor mavorixafor and nivolumab in advanced renal cell carcinoma patients with no prior response to nivolumab monotherapy. Invest New Drugs. 2021 Aug;39(4):1019-1027. doi: 10.1007/s10637-020-01058-2. Epub 2021 Jan 28. PMID 33507454

RESULTS

PARTICIPANT FLOW:
Groups:
- X4P-001 Plus Nivolumab: Participants received X4P-001 400 milligrams (mg) (as 4 capsules of 100 mg each) orally once daily in combination with nivolumab 240 mg intravenous (IV) infusion (over 60 minutes) every 2 weeks. Study medication was administered in 28-day cycles and continued until treatment-limiting toxicity or disease progression.
Period: Overall Study
Arm/Group | X4P-001 Plus Nivolumab
Started | 9
Received at Least 1 Dose of Study Medication | 9
Completed | 0
Not Completed | 9
Not completed — Adverse Event | 4
Not completed — Clinical Deterioration | 1
Not completed — Disease Progression | 3
Not completed — Study Termination | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study medication.
Groups:
- X4P-001 Plus Nivolumab: Participants received X4P-001 400 mg (as 4 capsules of 100 mg each) orally once daily in combination with nivolumab 240 mg IV infusion (over 60 minutes) every 2 weeks. Study medication was administered in 28-day cycles and continued until treatment-limiting toxicity or disease progression.
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Drug-related TEAEs: TEAEs with possible, probable, definite, or missing relationship to study medication (X4P-001 or Nivolumab). Serious AEs: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as events occurring on or after the first dose of study drug through 30 days after the last dose. Any TEAEs included both serious and non-serious TEAEs. A summary of other non-serious AEs and all serious AEs, regardless of causality, is located in Reported AE section.
Time Frame: From administration of first dose of study medication (Day 1) up to 30 days after last dose (up to 16 months)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 9
Participants
  Any TEAEs | 9
  Serious TEAEs | 2
  X4P-001-Related TEAEs | 9
  Nivolumab-Related TEAEs | 9

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of X4P-001
Description: Samples were to be analyzed for X4P-001 concentration using reversed-phase high performance liquid chromatography (RP-HPLC) with tandem mass spectrometry (MS) detection.
Time Frame: Predose (-30 minutes) on Day 1 of Cycle 1; predose (-10 minutes) on Days 8, 15, and 22 of Cycle 1, and Day 1 of Cycle 3; postdose at 60 and 90 minutes, and 2, 3 4, and 8 hours on Day 22 of Cycle 1
Population: The study was terminated and the pharmacokinetic (PK) samples collected could not be analyzed due to insufficient data available to assess the outcome measure as per the prespecified method of analysis.
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of X4P-001
Description: Samples were to be analyzed for X4P-001 concentration using RP-HPLC with tandem MS detection.
Time Frame: as for outcome 2
Population: The study was terminated and the PK samples collected could not be analyzed due to insufficient data available to assess the outcome measure as per the prespecified method of analysis.
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Minimum Plasma Concentration (Cmin) of X4P-001
Description: Samples were to be analyzed for X4P-001 concentration using RP-HPLC with tandem MS detection.
Time Frame: as for outcome 2
Population: as for outcome 3
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Reach Cmax (Tmax) of X4P-001
Description: Samples were to be analyzed for X4P-001 concentration using RP-HPLC with tandem MS detection.
Time Frame: as for outcome 2
Population: The study was terminated and the PK samples collected could not be analyzed due to insufficient data available to as per the prespecified method of analysis.
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With Objective Response, Evaluated Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR was defined as percentage of participants with best overall response of complete response (CR) or partial response (PR). CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) with a reduction in short axis to less than (<) 10 millimeters (mm). PR: At least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From administration of first dose of study medication (Day 1) until disease progression, study completion or early termination (up to 15 months)
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 9
percentage of participants | 11.1 [0.3 to 48.2]

7. Secondary Outcome: Duration of Objective Response (DOR), Evaluated Using RECIST Version 1.1
Description: DOR was defined as the time from first CR or PR whichever comes first until the time of disease progression by RECIST v1.1 or death due to any cause. CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) with a reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of 1 or more new lesions was also considered progression.
Time Frame: Time from first CR or PR until the time of disease progression or death due to any cause (up to 15 months)
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 9
months | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% confidence interval (CI) were not calculated.

8. Secondary Outcome: Time to Objective Response, Evaluated Using RECIST Version 1.1
Description: Time to objective response was defined as time from first administration of combination regimen to first CR or PR whichever comes first. CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) with a reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From administration of first dose of study medication (Day 1) until first appearance of CR or PR (up to 15 months)
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- X4P-001 Plus Nivolumab: Participants received X4P-001 400 mg (as 4 capsules of 100 mg each) orally once daily in combination with nivolumab 240 mg IV infusion (over 60 minutes) every 2 weeks. Study treatment was administered in 28-day cycles and continued until treatment-limiting toxicity or disease progression.
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 9
months | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI were not calculated.

9. Secondary Outcome: Disease Control Rate: Percentage of Participants With CR or PR or Stable Disease (SD), Evaluated Using RECIST Version 1.1
Description: Disease control rate was defined as percentage of participants with best overall response of CR or PR or SD. CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) with a reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of 1 or more new lesions was also considered progression.
Time Frame: as for outcome 6
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 9
percentage of participants | 88.9 [51.8 to 99.7]

10. Secondary Outcome: Progression Free Survival (PFS), Evaluated Using RECIST Version 1.1
Description: PFS was defined as the time from first administration of study medication until objective tumor progression or death from any cause. Tumor progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. An unequivocal progression of existing non-target lesions or the appearance of 1 or more new lesions was also considered progression.
Time Frame: From administration of first dose of study medication (Day 1) until disease progression or death from any cause (up to 15 months)
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 9
months | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI were not calculated.

11. Secondary Outcome: Time to Progression (TTP), Evaluated Using RECIST Version 1.1
Description: TTP was defined as the time from first administration of study medication until objective tumor progression. Tumor progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions or the appearance of 1 or more new lesions was also considered progression.
Time Frame: From administration of first dose of study medication (Day 1) until disease progression (up to 15 months)
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | X4P-001 Plus Nivolumab
Number analyzed (Participants) | 9
months | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI were not calculated.

ADVERSE EVENTS:
Time Frame: From administration of first dose of study medication (Day 1) up to 30 days after last dose (up to 16 months)
Description: Safety population included all participants who received at least 1 dose of study medication.
Arm/Group | X4P-001 Plus Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | X4P-001 Plus Nivolumab (N=9)
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Mucosal inflammation (General disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | X4P-001 Plus Nivolumab (N=9)
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Anal incontinence (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dry eye (Eye disorders) | 4
Conjunctival hyperaemia (Eye disorders) | 2
Lacrimation increased (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Weight decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Lipase increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 2
Chills (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Headache (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Ear congestion (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Bronchitis (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Due to low enrollment, the study was terminated early. Data for some pre-registered endpoints were therefore not collected or analysed and could not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT02923531/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02923531/SAP_001.pdf